CLINICAL TRIAL: NCT03942445
Title: In Vivo Analysis of Muscle Stem Cell Vascular Niche in Patients Presenting Chronic and Acute Lower Limb Ischemia (MyostemIschemia)
Brief Title: In Vivo Analysis of Muscle Stem Cells in Chronic and Acute Lower Limb Ischemia (MyostemIschemia)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C18-35
Record Dates: First submitted 2019-04-29; First posted 2019-05-08 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Artery Disease; Muscle Disorder
Keywords: Muscle ischemia; Satellite cells; Chronic limb ischemia; Endothelial cells
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All muscle biopsies are immediately labeled and routed to the lab where technicians and assessors are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control patients (Experimental)
  Interventions: Procedure: Gastrocnemius muscle biopsy
- Chronic ischemia (Experimental)
  Interventions: Procedure: Gastrocnemius muscle biopsy
- Acute ischemia (Experimental)
  Interventions: Procedure: Gastrocnemius muscle biopsy

INTERVENTIONS:
Procedure: Gastrocnemius muscle biopsy — In all groups, a 5 mm large gastrocnemius muscle biopsy will be performed and the samples immediately managed in experimental laboratory.

SUMMARY:
Skeletal muscle regenerates after injury, due to the satellite cells (SCs), the muscle stem cells that activate, proliferate, differentiate and fuse to form new myofibers. While SCs are indispensable for regeneration, there is increasing evidence for the need for an adequate cellular environment. Among the closest cellular partners of SCs are vascular cells. During muscle regeneration, endothelial cells (ECs) stimulate SC differentiation while SCs exhibit pro-angiogenic properties indicating a coupling between angiogenesis and myogenesis.The specific signaling cues controlling these relationships are still poorly characterized, specially in specific pathologic context such as limb ischemia. The investigators research aims to evaluate the role of chronic and acute lower limb ischemia on the SC status and interaction with ECs in human patients.

DETAILED DESCRIPTION:
Post-injury muscle regeneration is a multifaceted process requiring the coordination of myogenesis and angiogenesis. Whether this coordination is altered in pathological context has been poorly investigated, whether the original defect stems from the myogenic cell (degenerative myopathy) or the vessel (chronic limb ischemia).

Chronic limb ischemia in patients with peripheral arterial disease (PAD) causes muscle weakness and decreases exercise tolerance. PAD patients with chronic limb ischemia suffer mainly from intermittent claudication on walking or rest pain in more advanced stage, i.e. in critical limb ischemia . PAD is associated with muscle cell apoptosis and atrophy, fiber type switching (from type I to type II), increased muscle fat content and denervation . The underlying mechanisms are from hemodynamic origin and linked to atherosclerotic obstructions of the major arteries supplying the lower extremities. However, additional mechanisms contribute to the limb manifestations, where a reduction in blood flow alone cannot explain exercise limitation in symptomatic PAD patients. These mechanisms include a cascade of pathological responses during exercise-induced ischemia and reperfusion at rest, endothelial dysfunction, oxidative stress, inflammation, and muscle metabolic abnormalities). Surprisingly, the implication of SCs in the pathophysiology of chronic limb ischemia has been overlooked. One could assume that the regenerative capacity of SCs in advanced PAD is overwhelmed by prolonged ischemia. In this case, a decrease in SC regenerative capacities could participate in the aggravation of muscle atrophy and limb perfusion, considering their known pro-angiogenic properties. Consistently, a preclinical study demonstrated that combined delivery of pro-angiogenic and myogenic factors improves ischemic muscle recovery , while endovascular surgery and administration of angiogenic factors (recombinant proteins or gene therapy) or angiogenic cells (cell therapy) showed limited effects. This indicates that promoting angiogenesis along with myogenesis may be a more suitable therapeutic strategy.

Impaired angiogenesis and/or impaired myogenesis are thus novel players in chronic limb ischemia and could represent potential therapeutic targets to delay or alleviate muscle dysfunction.

For PAD patients, muscle biopsies will take place during femoro-popliteal bypass surgery. Control muscle biopsies will be performed in patients undergoing orthopedic surgery of the lower limb or femora-popliteal bypass for non-ischemic reasons (popliteal aneurysm, popliteal entrapment syndrome) In parallel, human SCs in non-PAD patients with <6h acute limb ischemia (from embolic origin) will be obtained. For the PAD study, patients with autoimmune disease, active cancer, end stage renal disease or tissue necrosis or edema close to the site of biopsy will be excluded from this study.

Three major assessments will be performed:

1. Topographic study: Number, distribution, and relative proximity of SC, and capillaries, fiber type, based on immunohistochemistry applied to standard thin transverse sections, and to thicker segments of cleared muscle.
2. Functional study: in vitro and in vivo comparison of myogenic potential of SC between ischemic and control patients, based on SC primary cell culture, and SC-ECs co-culture system. Ultimately, SC transplantation in injured muscle of immunodepressed mice will aim to evaluate myogenic capacities.
3. Transcriptomic analysis: of SCs and ECs sorted from ischemic muscle from PAD patients, control muscle and patients with acute ischemia.

The investigators goal is to analyze and compare the molecular adaptation of ECs and SCs towards chronic ischemia (in a context of muscle atrophy and weakness) as compared with acute ischemia (in a context of normal muscle function) Particular attention in the analysis will be given to the pathways already involved in myogenesis/angiogenesis coupling during muscle regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Non PAD patients undergoing vascular surgery for non-occlusive lesions or undergoing orthopedic surgery with gastrocnemius muscle exposure
* PAD patients > Rutherford Stage 3 or with Chronic Threatening Limb Ischemia, undergoing vascular surgery with gastrocnemius muscle exposure
* Patients presenting acute limb ischemia and undergoing vascular surgery with gastrocnemius muscle exposure

Exclusion Criteria:

* Major Limb edema
* Muscle necrosis
* Acute on chronic ischemia
* Auto-immune vasculitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Differential expression of genes involved in myogenesis and angiogenesis | April 2019 - October 2021
  Transcriptomic study through RNA Seq

SECONDARY OUTCOMES:
Comparative study of the topography of SC and ECs | April 2019 - October 2021
  Number of SC, capillaries, distance to each others, fiber type, number and diameter of muscle fibers
Comparative study of myogenic capacity: In vitro differentiation of SC during primary cell culture | April 2019 - October 2021
  Number of induced myotubes, shape of myotubes, presence of myonuclei (Score 0: Normal, 1: Dystrophic) during cell culture:
In vitro comparative study of angiogenic capacity | April 2019 - October 2021
  Number of induced vessels in a co-culture system (SC/HUVECs)
Myogenic and Angiogenic capacity of transplanted SC (in mice tibialis anterior) | April 2019 - October 2021
  Ability to induce muscle regeneration, revascularisation, and SC original pool renewal:
  Measurements performed at day 0, 5, 7, 14, 21 days after SC transplantation and tibias anterior lesion
  * Evolution of the number of SC per 100 myofibers
  * Evolution of the number of capillaries per 100 myofibers
  * Evolution of the myofibers diameter
  * Surface of necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Touma, Dr, Principal Investigator — Hôpital Henri Mondor, service de chirurgie vasculaire, 51 avenue Maréchal de Lattre de Tassigny, 94010 Créteil
Locations (1):
- Hôpital Henri Mondor, service de chirurgie vasculaire, 51 avenue Maréchal de Lattre de Tassigny, 94010 Créteil, Paris, France

IPD SHARING:
Plan to Share IPD: No